CLINICAL TRIAL: NCT01190345
Title: Phase II" Proof of Concept " Trial Evaluating Anti Cancer Stem Cell Activity of Pre-operative Bevacizumab in Combination With Chemotherapy in Breast Cancer
Brief Title: Anti Cancer Stem Cell Activity of Pre-operative Bevacizumab and Chemotherapy in Breast Cancer
Acronym: AVASTEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVASTEM/IPC 2009-001
Record Dates: First submitted 2010-08-24; First posted 2010-08-27 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WITH bevacizumab (Experimental): bevacizumab 15 mg/kg on day 1 of each cycle : 4 cycles of 5-fluorouracil 500 mg/m² IV + epirubicin 100 mg/m² IV + cyclophosphamide 500 mg/m² IV (FEC100) every 21 days and 4 cycles of docetaxel 100 mg/m² IV every 21 days.
  Patients with HER2+ disease will receive trastuzumab (8 mg/kg (IV then 6 mg/kg, every 21 days), which will be started with docetaxel and administered for a total duration of 54 weeks, 18 injections.
  Interventions: Drug: bevacizumab
- without bevacizumab (Active Comparator): 4 cycles 5-fluorouracil 500 mg/m² IV + epirubicin 100 mg/m² IV + cyclophosphamide 500 mg/m² IV of (FEC100) every 21 days and 4 cycles of docetaxel 100 mg/m² IV every 21 days.
  Patients with HER2+ disease will receive trastuzumab (8 mg/kg (IV then 6 mg/kg, every 21 days), which will be started with docetaxel and administered for a total duration of 54 weeks, 18 injections.
  Interventions: Drug: no bevacizumab

INTERVENTIONS:
Drug: bevacizumab — Patients receive on day 1 of each cycle : bevacizumab 15 mg/kg (8 injections in total).
  Other Names: avastin
  Arms: WITH bevacizumab
Drug: no bevacizumab — no bevacizumab
  Arms: without bevacizumab

SUMMARY:
The purpose of this study is to evaluate anti-cancer stem cell (CSC) activity (measured by the amount of Aldehyde dehydrogenase 1/ALDH1+ cells before and after treatment) of pre-operative bevacizumab in combination with conventional chemotherapy in breast cancer receiving neo-adjuvant treatment, compared to a control arm receiving chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 ys
* Primary breast cancer treated in the neoadjuvant setting (synchronous metastatic disease are eligible)
* Primary breast tumor accessible to initial biopsy
* White Blood Count > 3.000/µl and Absolute neutrophil count ≥ 1.500/µl AND platelets ≥ 100 x 109/L AND Hemoglobin ≥ 9 g/dL, Serum creatinine ≤ 150µm/l• Urine dipstick for proteinuria < 2+. Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours, Total bilirubin ≤ 1.5 ULN and ASAT < 2.5 ULN AND ALAT < 1.5 ULN (2.5 if liver metastasis), Adequate coagulation function: International normalized ratio (INR) ≤ 1.5 and TCA ≤ 1.5 x ULN
* Left ventricular ejection fraction (LVEF) ≥ 55% (isotopic or
* ultrasound methods)
* Karnofsky Index > 1 ; Performance status 0 to 1
* Patients must have signed a written informed consent form prior to any study specific screening procedures
* Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen.

Exclusion Criteria:

* Previous history of cancer (other than curatively treated basal and squamous cell carcinoma of the skin and/or in-situ carcinoma of the cervix) relapsing within the 5 years before study entry
* Known contra-indication to anticancer compounds used
* Uncontrolled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg) or history of hypertensive encephalopathy
* History of inherited diathesis or recent thrombotic events
* Non-healing wound, active peptic ulcer or bone fracture.
* Major surgery or significant traumatic injury within 28 days prior to study treatment start
* History of abdominal fistula, trachea-oesophageal fistula or urinary fistula
* Use of Non Steroid Anti Inflammatory or full dose anticoagulants or antiaggregation treatments within 10 days
* Pregnancy and breast feeding, premenopausal patient and no effective contraception
* Brain metastasis.
* Any unstable severe disease such as : uncontrolled cardiac or vascular disease, uncontrolled hemorrhagy, uncontrolled neuropsychiatric disorders, including dementia, uncontrolled infection or any severe disorders that may preclude study participation
* Patient considered geographically, socially or psychologically unable to comply with the treatment and the required medical follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-05 (Actual); Primary Completion 2012-07-24 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Measure of the anti-cancer stem cell activity | 4 months
  The anti-cancer stem cell (CSC) activity is measured by the amount of Aldehyde dehydrogenase 1/ALDH1+ cells after 4 cycles of treatment compared to the amount before treatment

SECONDARY OUTCOMES:
Evaluation of the safety of the treatment | 8 months
  Evaluation of the safety of the treatment at each cycle, estimated by the number of patients with clinical and biological adverse events coded according to the CTCAE
Evaluation of the disease-free survival, recurrence-free survival and overall survival | 5 years
  The disease-free survival, recurrence-free survival and overall survival are calculated from the inclusion to the time of the event
Evaluation of the pathological complete response rate | 8 months
  Evaluation of the pathological complete response rate according to the classification of Sataloff

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc EXTRA, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (3):
- France (3):
  - Jean-Marc EXTRA, MD, Marseille
  - Jean-Yves PIERGA, Paris
  - Hervé CURE, Reims

REFERENCES:
- See also: institut Paoli-Calmettes web site — http://www.institutpaolicalmettes.fr/